CLINICAL TRIAL: NCT04804046
Title: Defining Microbial and Immune Changes Following Synbiotic Supplementation in Post-operative Crohn's Disease Patients
Brief Title: Synbiotics and Post-op Crohn's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Alberta (Other)
Collaborators: W. Garfield Weston Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00092967
Record Dates: First submitted 2021-03-11; First posted 2021-03-18 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Inflammation; Probiotics; Prebiotics; Dietary Fiber; Synbiotics; Gut Microbiome
MeSH Terms: conditions — Crohn Disease; Inflammation | interventions — Synbiotics; arabinoxylan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic (Experimental): Bifidobacterium longum spp. longum R0175, Bifidobacterium animalis spp. Lafti B94, Bifidobacterium bifidum R0071 at 3x10^9 CFU/d plus resistant starch type 2, arabinoxylan, and galactooligosaccharide at 24 g/d will serve as the treatment.
  Interventions: Dietary Supplement: Synbiotic
- Digestible Maltodextrin (Placebo Comparator): Digestible maltodextrin will serve as the placebo.
  Interventions: Other: Digestible Maltodextrin

INTERVENTIONS:
Dietary Supplement: Synbiotic — Eighteen participants with Crohn's disease that are undergoing an ileocecal resection will supplement their normal diet with three Bifidobacterium spp. (3x10^9 CFU) plus three dietary fibers (24 g fiber) daily for six months.
  Other Names: Resistant starch type 2; HiMaize 260; Ingredion; Arabinoxylan; Naxus; Bioactive; Galactooligosaccharide; Vivinal; FrieslandCampina
  Arms: Synbiotic
Other: Digestible Maltodextrin — Eighteen participants with Crohn's disease that are undergoing an ileocecal resection will supplement their normal diet with Maltodextrin daily for six months.
  Other Names: Maltodextrin GLOBE Plus 15; Ingredion
  Arms: Digestible Maltodextrin

SUMMARY:
Crohn's disease (CD) is a lifelong incurable condition that causes inflammation of the intestinal tract of humans. The exact cause of CD is unknown, but genetics, diet, and the gut microbiome are all thought to play a major role. Many patients with CD will require surgery to remove affected portions of the gut, with ileocecal resections being the most common procedure performed. Regrettably, there is up to an 85% chance that disease returns to the surgical site. Strong immune suppressive medications may help to prevent disease relapse. However, patients are then at risk of serious side effects. Currently, no ideal post-op care exists for CD patients.

This study aims to assess whether a post-op synbiotic therapy (i.e. probiotics plus dietary fiber) prevents disease relapse in participants with CD. To test this, participants will consume probiotics (strains of bifidobacteria) before their surgery and then probiotics plus fiber supplements after surgery. Probiotics are live bacteria that have been shown to reduce inflammation of the gut. Fiber is given after surgery to help promote beneficial bacterial taxa and prevent less favorable bacterial taxa from triggering CD relapse. Patients will take the supplements for 6 months following surgery. They will be seen monthly to assess the effects of treatment on quality of life, symptoms of disease recurrence, inflammatory markers, and the gut microbiome. All patients will also undergo a colonoscopy at the end of the study to check for endoscopic reoccurrence.

DETAILED DESCRIPTION:
Crohn's disease (CD) is characterized by chronic intestinal inflammation and commonly involves the ileocecal region. Due to disease complications, many patients with CD require an ileocecal resection (ICR). However, disease often recurs postoperatively at the surgical anastomosis, with endoscopic recurrence rates as high as 85%. While the immunosuppressant infliximab has been shown to reduce endoscopic disease recurrence, it was not shown to prevent clinical relapse. The timing of infliximab treatment might be critical, as starting infliximab immediately after surgery rather than at the time of post-surgical recurrence resulted in 1-year remission rates of 92% and 57%, respectively. Currently, no ideal postoperative care exists for patients with CD. Thus, new approaches are required.

The gut microbiome has long been thought to play a causative role in the high rates of CD recurrence following surgical resection. Immediately following ICR, a state of inflammation and oxidative stress promotes aerotolerant microbes at the expense of beneficial short-chain fatty acid (SCFA)-producing anaerobes. The mucosal microbial composition in CD patients at the time of surgery is predictive of future disease relapse. Specifically, patients with a dominance of SCFA-producing anaerobic bacteria in the ileal mucosa at the time of surgical resection are more likely to remain in remission compared with patients which have a dominance of aerotolerant bacteria. Nutritional adjuncts based on probiotics or prebiotics could be applied to shift gut microbial imbalances towards SCFA-producers.

Though research is limited, probiotics containing bifidobacteria but not lactobacilli have been shown to lessen mucosal inflammation and recurrence rates when provided immediately post ICR. In a previous clinical trial, it was found that patients with CD that started the probiotic VSL#3 (4 Lactobacillus; 3 Bifidobacterium; 1 Streptococcus strains) immediately post surgery had reduced mucosal inflammatory cytokines and lower recurrence rates when compared to patients that started VSL#3 at 3-months post surgery. A smaller trial using VSL#3 in combination with antibiotic treatment also showed lower rates of endoscopic recurrence at 3- and 12-months following surgery. These results suggest that probiotic composition and treatment timing are critical for efficacy. While synergy between probiotics and prebiotics might improve clinical effects, the efficacy of synergistic synbiotics remains unknown. The aims of this study are the following:

AIM 1. Perform a parallel two-arm, randomized controlled exploratory trial in CD patients undergoing ICR to determine the safety and tolerability of a synbiotic treatment.

This is a pilot study in patients with CD undergoing ileocecal resection to evaluate the feasibility of supplementation with a synbiotic preparation that contains a mixture of resistant starch type 2 (HiMaize 260; Ingredion), arabinoxylan (Naxus; Bioactive), and galactooligosaccharide (Vivinal; FrieslandCampina) (24g/d) fibers plus probiotic bacteria (Bifidobacterium longum spp. longum R0175, Bifidobacterium animalis spp. Lafti B94, Bifidobacterium bifidum R0071; Lallemand Health Solutions) (3x10^9 CFU/d). Participants will be given the probiotics 2 days prior to surgery and then the synbiotic will both be given 7 days after surgery and will be consumed daily for 6 months. Digestible maltodextrin will be used as a placebo control (Maltodextrin GLOBE Plus 15; Ingredion). A total of 36 volunteers will be enrolled, stratified by sex, and randomized to one of 2 groups via computer-generated numbers, as well as blinded to their group allocation to reduce bias. Safety and tolerability of synbiotic (primary outcome) will be determined by the percentage of participants who experience treatment emergent adverse events and serious adverse events. Symptom and quality of life questionnaires will also be used to evaluate tolerance.

AIM 2. Determine if synbiotic therapy attenuates mucosal and systemic inflammation and reduces rates of disease relapse.

Each month, clinical recurrence will be evaluated by Harvey Bradshaw Index and C-reactive protein, serum cytokines (TNF-α, IL-6, IL-8, and IL-10), intestinal barrier markers (LPS, LPS-binding protein, and zonulin), and fecal calprotectin levels will be measured. At 6-months, endoscopic recurrence will be determined by Rutgeerts Index and biopsies will be taken for the assessment of mucosal inflammation.

AIM 3. Evaluate the impact on compositional and functional features of the fecal microbiota and to characterize associations between clinical and microbial outcomes.

Fecal samples will be collected each month for the characterization of the microbiota by 16S rRNA gene sequencing. Fecal concentrations of SCFAs and bile acids will also be determined as functional measures of the gut microbiota. Associations between clinical outcomes and microbiota features will be assessed to identify signatures that predict the synbiotic impact.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease
* Undergoing ileocolonic resection
* Females of childbearing potential must agree to use a medically approved method of birth control (e.g. hormonal contraception, intrauterine devices, vasectomy/tubal ligation, barrier methods, double-barrier method) and must have negative pregnancy test results at screening and baseline.

Exclusion Criteria:

* Subjects which are reliant on partial or total parenteral nutrition
* Subjects with permanent or temporary diverting ileostomies
* Subjects with gluten intolerance/sensitivity
* Subjects with milk or soy allergy
* Subjects with diabetes, immune disorders, or bleeding disorders
* Subjects with any documented psychological disorders
* Pregnant women, women who are breast feeding, or women planning on becoming pregnant
* Subjects with perforation or ischemia of the gut
* Subjects unable to tolerate any oral intake following surgery
* Subjects with immune-compromised condition (e.g. AIDS, lymphoma)
* Subjects who are taking tetracycline
* Subjects with uncontrolled cardiovascular or respiratory disease or active malignancy
* Subjects who are enrolled in another clinical trial
* Subjects who are unable to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The percentage of participants who experience treatment emergent adverse and serious adverse events | 6-month period
  The primary objective of this study is to determine the safety and tolerability of a synbiotic treatment as assessed by the percentage of participants who experience treatment emergent adverse and serious adverse events.

SECONDARY OUTCOMES:
Changes in quality of life (1) | 6-month period
  Synbiotic induced changes in quality of life as assessed by the EQ-ED5 at baseline and 6 months.
Changes in quality of life (2) | 6-month period
  Synbiotic induced changes in quality of life as assessed by the Short Inflammatory Bowel Disease Questionnaire between baseline and 6 months.
Prevention of clinical recurrence | 6-month period
  Clinical recurrence will be defined as Harvey Bradshaw index >5 at 6 months
Prevention of endoscopic recurrence | 6-month period
  Endoscopic recurrence will be defined as >2 Rutgeerts score at 6 months
Changes in systemic inflammation | 6-month period
  Synbiotic induced changes in systemic inflammation (CRP, TNF-α, IL-6, IL-8, and IL-10), will be assessed between baseline and 6 months.
Changes in intestinal inflammation | 6-month period
  Synbiotic induced changes in intestinal inflammation (fecal calprotectin) will be assessed between baseline and 6 months.
Changes in intestinal barrier function | 6-month period
  Synbiotic induced changes in intestinal barrier function (LPS, LPS-binding protein, and zonulin) measures will be assessed between baseline and 6 months.
Changes in the fecal microbiota composition | 6-month period
  Synbiotic induced changes in microbial composition by 16S rRNA gene sequencing will be assessed at baseline and 6 months.
Changes in fecal short chain fatty acids | 6-month period
  Synbiotic induced changes in the levels of SCFAs in fecal samples will be assessed between baseline and 6 months.
Changes in fecal bile acids | 6-month period
  Synbiotic induced changes in fecal bile acids will be assessed between baseline and 6 months.
Time to first bowel movement | Immediately post-surgery up to 7 days
  Probiotic induced changes in the time to the participant's first bowel movement will be recorded.
Time to hospital discharge | Post-surgery up to 30 days
  Probiotic induced changes in the time to the participant's to hospital discharge will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Madsen, PhD, Principal Investigator — University of Alberta
Locations (5):
- Canada (5):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - University of Alberta Human Nutrition Research Unit, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No